CLINICAL TRIAL: NCT05478668
Title: Predictors of Pain Chronicity in Patients With Gunshot and Mine-explosive Wounds
Acronym: PPСPGM-EW
Status: Completed | Type: Observational
Sponsor: Bogomolets National Medical University (Other)
Responsible Party: Principal Investigator, Vasyl' Horoshko, I am obtaining the scientific degree of Doctor of Medical Sciences at the Department of Surgery, Anesthesiology and Intensive Care, Bogomolets National Medical University
Other Study IDs: №158, 2022.23.05
Record Dates: First submitted 2022-07-26; First posted 2022-07-28 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: Chronic Pain, Widespread
Keywords: Chronic pain, gunshot wounds, mine-explosive wounds
MeSH Terms: conditions — Chronic Pain; Wounds, Gunshot

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- retrospective analysis: A retrospective analysis of disease histories for the period from 2014 to 2021 was carried out. Data collection was carried out at all stages of treatment: medical and nursing brigade, military mobile hospital, military medical clinical center, during rehabilitation, within 12 months of the injury. In all patients, the assessment of anesthetic risk was carried out according to the ASA scale. The basic tool for pain intensity research was a visual analog scale. Intervals between analgesia were also studied. The study of the neuropathic component of pain was carried out using the Didier Bouhassiraa neuropathic pain diagnostic questionnaire. Study of the presence of an acute stress reaction scale The Hospital Anxiety and Depression Scale. Research on the presence of post-traumatic stress disorders was carried out using the Mississippi scale of post-traumatic stress disorders (military version). Satisfaction with treatment results was studied using the Chaban Quality of Life Scale.
  Interventions: Other: visual analog scale
- prospective study: Recruitment of patients for the prospective study was carried out in the period from 02.24.2022 to 05.24.2022. Data collection was carried out during the Russian invasion of Ukraine and the offensive on Kyiv. All patients with gunshot wounds were evacuated to the stage of treatment - the National Military Medical Clinical Center "Main Military Clinical Hospital". The research was conducted using the same methods as during the retrospective analysis. The exception was the study period during treatment at the military medical clinical center: here it was 14 days.
  Interventions: Other: visual analog scale

INTERVENTIONS:
Other: visual analog scale — In all patients, the assessment of anesthetic risk was carried out according to the ASA scale. The basic tool for pain intensity research was a visual analog scale. Intervals between analgesia were also studied. The study of the neuropathic component of pain was carried out using the Didier Bouhassiraa neuropathic pain diagnostic questionnaire. Study of the presence of an acute stress reaction The Hospital Anxiety and Depression Scale. Research on the presence of post-traumatic stress disorders was carried out using the Mississippi scale of post-traumatic stress disorders (military version). Satisfaction with treatment results was studied using the Chaban Quality of Life Scale.
  Other Names: neuropathic pain Didier Bouhassiraa, Nadine Attala et al. Pain, 2005, 114: 29-36 (DN4).; Chaban Quality of Life Scale; The Hospital Anxiety and Depression Scale; Mississippi scale of post-traumatic stress disorders (military version) (MS PTSD (m))

SUMMARY:
82.1% of patients with gunshot and mine-explosive wounds during hostilities in Ukraine have negative results of pain treatment, which leads to its chronicity. Identifying predictors of pain chronicity in these patients may improve their treatment outcomes.

DETAILED DESCRIPTION:
The study of predictors of pain chronicity in patients with gunshot and mine-explosive wounds requires in-depth study, because the subjective feelings and emotional experiences experienced by patients during the wounding in combat conditions have their own characteristics. Since pain becomes chronic in 82.1%, the data of our study will play an important role in preventing the chronicity of pain.

ELIGIBILITY:
Inclusion Criteria:

* the presence of gunshot and mine-explosive injuries

Exclusion Criteria:

* absence of gunshot and mine-explosive injuries

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study was carried out on the basis of the National Military Medical Clinical Center "Main Military Clinical Hospital". All patients participated in Operation Joint Forces and received gunshot wounds during combat operations.
  A retrospective analysis of disease histories for the period from 2014 to 2021 was carried out. Data collection was carried out at all stages of treatment: medical and nursing brigade, military mobile hospital, military medical clinical center, during rehabilitation, within 12 months of the injury.
  Recruitment of patients for the prospective study was carried out in the period from 02.24.2022 to 05.24.2022. Data collection was carried out during the Russian invasion of Ukraine and the offensive on Kyiv.
Sampling Method: Non-Probability Sample
Enrollment: 2215 (Actual)
Dates: Start 2022-02-24 (Actual); Primary Completion 2022-05-24 (Actual); Study Completion 2022-05-24 (Actual)

PRIMARY OUTCOMES:
visual analog scale | 1 year
  evaluation of the number of points
Didier Bouhassiraa DN4 | 1 year
  evaluation of the number of points
The Hospital Anxiety and Depression Scale | 1 year
  evaluation of the number of points
Chaban Quality of Life Scale | 1 year
  evaluation of the number of points
Mississippi PTSD scale (military version) | 1 year
  evaluation of the number of points

CONTACTS AND LOCATIONS:
Locations (1):
- Bogomolets National Medical University, Ministry of Health of Ukraine, Kyiv, Ukraine

IPD SHARING:
Plan to Share IPD: Undecided
I plan to share